CLINICAL TRIAL: NCT01546350
Title: Comparison of Standard ART Practice vs. Trophectoderm Biopsy, Array CGH Analysis, and Day-6 Replacement of a Single Euploid Embryo
Brief Title: Preimplantation Genetic Diagnosis Using Blastocyst Biopsy and Array CGH
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: not enough patients recruited on time
Sponsor: Reprogenetics (Industry)
Collaborators: Reprogenetics, Livingston, NJ (Unknown); Long Island IVF, Melville, NY (Unknown); Reproductive Associates of Illinois, Highland Park, IL (Unknown); Yale University (Other); McGill University (Other); BlueGnome, Cambridge, UK (Unknown); Southern California Reproductive Center, CA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Reprogenetics study 389; Reprogenetics study 389 (Other: Reprogenetics)
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-05

CONDITIONS: Infertility; Recurrent Pregnancy Loss
Keywords: infertility, recurrent pregnancy loss, miscarriage
MeSH Terms: conditions — Infertility; Abortion, Spontaneous | interventions — Prostaglandins D

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control - regular ART treatment (No Intervention): patients will have up to two embryos replaced on day 5 based on morphological and developmental characteristics, and the other embryos reaching blastocyst stage will be vitrified. If patients in the control group do not have a pregnancy to term from that fresh cycle, they will be offered free PGD either for the frozen embryos of that cycle or for the next cycle (up to the center and patient). Data from that PGD is not part of the study.
- Test - PGD (Experimental): patients will have grade A,B or C blastocysts hatched on day 5, biopsied on day 5, analyzed by array CGH, and a single euploid embryo transferred on day 6. Any morulas developing to grade A,B or C blastocyst on day-6 will be also analyzed but vitrified for use in a future cycle.
  Interventions: Genetic: PGD; Procedure: PGD

INTERVENTIONS:
Genetic: PGD — array CGH after blastocyst biopsy
  Other Names: PGD: Preimplantation Genetic Diagnosis
  Arms: Test - PGD
Procedure: PGD — PGD using blastocyst biopsy and testing of the biopsy by array CGH
  Arms: Test - PGD

SUMMARY:
The investigators propose to perform a clinical randomized trial to evaluate the effect of single embryo (blastocyst) transfer (SET) with array CGH for the evaluation of the complete chromosome complement of the blastocyst in comparison to standard ART methods in which one or more embryo are replaced. Patients will be randomized into two groups:

* Control group: patients will have up to two embryos replaced on day 5 based on morphological and developmental characteristics, and the other embryos reaching blastocyst stage will be vitrified. If patients in the control group do not have a pregnancy to term from that fresh cycle, they will be offered free PGD either for the frozen embryos of that cycle or for the next cycle (up to the center and patient). Data from that PGD is not part of the study.
* Test group: patients will have grade A,B or C blastocysts hatched on day 5, biopsied on day 5, analyzed by array CGH, and a single euploid embryo transferred on day 6. Any morulas developing to grade A,B or C blastocyst on day-6 will be also analyzed but vitrified for use in a future cycle.

DETAILED DESCRIPTION:
Patients will be randomized after fertilization, and will be dropped from the study if they produce 3 or less blastocysts on day 5. The Primary efficacy endpoint of comparing the study group with the control will be (I) implantation rates and (II) multiple pregnancies (twin or higher order) comparing the first transfer.

The study may be extended to evaluate secondary efficacy endpoints which will be miscarriage rate and take home baby rates comparing the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age 33 to 42 years old (included)

Exclusion Criteria:

* MESA and TESE patients
* At least one partner carrier of a chromosomal or genetic disease
* Abnormal ovarian reserve, defined as FSH of >10 IU/L on day 2-4 of the cycle and AMH < 1ng /ml (If only one of the two parameters altered then patients is acceptable).
* Egg donor cycle (sperm donor is acceptable)

Exclusion criteria during stimulation:

* Less than eight antral follicles on day 2-4 of cycle

Exclusion criteria on day 5 post retrieval:

* Patients will be excluded if they produce less than 3 grade A,B or C blastocysts by day 5.

Ages: 32 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | First month after replacement
  fetal sacs / embryos replaced

SECONDARY OUTCOMES:
Spontaneous miscarriage rate | during first and second trimester of pregnancy
  pregnancies lost / pregnancies of cycles randomized
ongoing pregnancy rate | third trimester of pregnancy
  pregnancies past second trimester / cycles started
Multiple pregnancy rate | first month after transfer
  Twin or multiple order pregnancies / total pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Munne, PhD, Study Director — Reprogenetics
Locations (4):
- United States (4):
  - Southern California Reproductive Center, Beverly Hills, California
  - Reproductive Associates of Illinois, Highland Park, Illinois
  - Reprogenetics, Livingston, New Jersey
  - Long Island IVF, Melville, New York

REFERENCES:
- [Background] Gutierrez-Mateo C, Colls P, Sanchez-Garcia J, Escudero T, Prates R, Ketterson K, Wells D, Munne S. Validation of microarray comparative genomic hybridization for comprehensive chromosome analysis of embryos. Fertil Steril. 2011 Mar 1;95(3):953-8. doi: 10.1016/j.fertnstert.2010.09.010. Epub 2010 Oct 25. PMID 20971462
- [Background] Cohen J, Wells D, Munne S. Removal of 2 cells from cleavage stage embryos is likely to reduce the efficacy of chromosomal tests that are used to enhance implantation rates. Fertil Steril. 2007 Mar;87(3):496-503. doi: 10.1016/j.fertnstert.2006.07.1516. Epub 2006 Dec 4. PMID 17141767
- [Background] Munne S, Wells D, Cohen J. Technology requirements for preimplantation genetic diagnosis to improve assisted reproduction outcomes. Fertil Steril. 2010 Jul;94(2):408-30. doi: 10.1016/j.fertnstert.2009.02.091. Epub 2009 May 5. PMID 19409550
- [Background] Schoolcraft WB, Fragouli E, Stevens J, Munne S, Katz-Jaffe MG, Wells D. Clinical application of comprehensive chromosomal screening at the blastocyst stage. Fertil Steril. 2010 Oct;94(5):1700-6. doi: 10.1016/j.fertnstert.2009.10.015. Epub 2009 Nov 25. PMID 19939370
- [Background] De Vos A, Staessen C, De Rycke M, Verpoest W, Haentjens P, Devroey P, Liebaers I, Van de Velde H. Impact of cleavage-stage embryo biopsy in view of PGD on human blastocyst implantation: a prospective cohort of single embryo transfers. Hum Reprod. 2009 Dec;24(12):2988-96. doi: 10.1093/humrep/dep251. Epub 2009 Sep 21. PMID 19773223